CLINICAL TRIAL: NCT01669876
Title: 3-Month, Single Site or Multi-Site, Double Blind, Randomized, Placebo-Controlled, Parallel-Group Trial to Evaluate the Safety Tolerability and Potential Effects of the Dietary Supplement Anatabloc(R) in Subjects With Alzheimer's Disease
Brief Title: Study to Evaluate Dietary Supplementation With a Version of Anatabloc(R) in Subjects With Alzheimer's Disease
Acronym: ASAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative status of active ingredient anatabine
Sponsor: Rock Creek Pharmaceuticals, Inc. (Industry)
Collaborators: Roskamp Institute Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCP-009
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Alzheimer Disease
Keywords: Randomized; Double-Blind; Dietary Supplements
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement: Anatabloc(R) (Active Comparator): Study product, as mint-flavored lozenge (3 mg anatabine per lozenge) to be taken 2-3 times each day
  Interventions: Dietary Supplement: Anatabloc(R)
- Placebo (Placebo Comparator): Placebo, as mint-flavored lozenge, to be taken 2-3 times each day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Anatabloc(R) — Dietary supplement Anatabloc(R), as a mint-flavored lozenge, to be taken 2-3 times each day
  Arms: Dietary Supplement: Anatabloc(R)
Dietary Supplement: Placebo — Placebo, as a mint-flavored lozenge, to be taken 2-3 times each day
  Arms: Placebo

SUMMARY:
To explore whether dietary supplementation with a version of Anatabloc(R) exerts an effect on blood levels of amyloid beta (Aβ), or impacts global or functional measures of Alzheimer's Disease (AD) in subjects with mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old.
* Have a diagnosis of probable AD or a concurrent diagnosis of probable AD and possible or probable vascular dementia.
* Score 16 or more on the Mini-Mental State Examination (MMSE).
* Otherwise stable medical history and general health.
* Weigh between 45 kg and 120 kg inclusive.

Exclusion Criteria:

* Have contra-indications, allergy, or sensitivity to the study products or their components.
* Be currently taking any of the following medications: systemic (oral or injectable) glucocorticoids; interferon-alpha; anti-CD20 antibody (e.g., rituximab); or anti-CTLA-4 antibody (e.g., ipilimumab).
* Be a current smoker or smokeless tobacco user.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse effects when using the supplement | 3 months
  Collected data on the numbers and types of adverse effects among subject individuals with mild to moderate Alzheimer's disease (AD).

SECONDARY OUTCOMES:
Measured changes in blood markers of AD | 3 months
  Changes in blood levels of amyloid beta (Aβ)
Changes in global or functional measures of AD in subjects during the course of the study | 3 months
  Changes in subject's scores in global and functional measures of AD during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: A Keegan, MD, Principal Investigator — Roskamp Institute
Locations (1):
- Roskamp Institute, Sarasota, Florida, United States